CLINICAL TRIAL: NCT06982833
Title: Investigation of the Effect of Trunk Restraint on Upper Extremity Functionality in Individuals With Multiple Sclerosis
Brief Title: Trunk Restraint in Multiple Sclerosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zonguldak Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, ARZUCAN TOKSAL UÇAR, PhD, Zonguldak Bulent Ecevit University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Trunk Restraint
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Multiple Sclerosis; Healthy Control
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: MS patients and their age-matched healthy control group were evaluated.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Multiple Sclerosis (Experimental): Patients and healthy individuals first filled out the demographic and clinical information form. Then, the Trunk Impairment Scale was evaluated. Participants performed 9DPT with their trunks free and again with their trunks restrained.
  Interventions: Other: Trunk restraint

INTERVENTIONS:
Other: Trunk restraint — Participants were seated in a chair with a standard sitting height of 26 centimeters. After completing the 9-Hole Peg Test with their trunks free on a table of appropriate height so that their trunks would not flexion, they were secured to the chair crosswise in front of their chest with the help of a non-elastic but firm enough belt that would not cause discomfort to the person. Participants completed the 9-DPT with their trunks constrained.

SUMMARY:
This study examined the effect of trunk restraint on upper extremity functionality in patients with Multiple Sclerosis (MS).The study included 66 MS patients over the age of 18 and 30 healthy individuals. Participants' upper extremity functions were assessed. Their trunks were then restrained and their upper extremity functions were assessed again. The patients' level of disability (EDSS), trunk control (Trunk Impairment Scale - TIS), upper extremity functionality (Nine Hole Peg Test- 9HPT), were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Being over 18 years old
* Being diagnosed with MS
* Volunteering

Exclusion Criteria:

* Having any additional disease or disorder of the upper extremity or trunk (such as disc herniation, fracture)
* Having any additional neurological disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-04-10 (Actual); Study Completion 2025-04-15 (Actual)

PRIMARY OUTCOMES:
Expanded Disability Status Scale (EDSS) | up to 6 weeks
  EDSS was used to determine the patients' level of disability. EDSS is most commonly used to assess the level of disability in persons with MS. In this scale pyramidal, cerebral, cerebellar, brainstem, visual and sensory subparameters are evaluated it consists of ordinal rating system ranging from 0 (normal neurological status) to 10 (death due to MS) in 0.5 increments interval (when reaching EDSS 1). The lower scale values of the EDSS measureimpairments based on the neurological examination, while the upper range of the scale (> EDSS 6) measures handicaps of patients with MS. The determination of EDSS 4 - 6 is heavily dependent on aspects of walking ability.
Trunk Impairment Scale (TIS) | up to 6 weeks
  This scale used to evaluate the trunk control of the participants, TIS contains static sitting balance, dynamic sitting balance, and coordination. The total score of this scale is from 0 to 23 and a high score indicates better trunk control.
  The patients were placed in the standard sitting position for the test and the parameters were applied. Standart position is such that the knees are flexed at 90 degrees, without back support, with the hands and forearms on the thighs and the feet in contact with the ground.
Nine-Hole Peg Test (9HPT) | up to 6 weeks
  It is a short, standardized, quantitative test used to evaluate upper extremity function. In the test, patients are asked to pick up nine wooden pegs from a platform as quickly as possible and then place them back into the holes.In our study, the test was conducted twice for both the dominant and non-dominant hands, and the average completion time was recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Güngör Beyza Özvar Şenöz, PhD, Principal Investigator — Yuksek Ihtisas University; Bilge Piri Çınar, Assoc. Prof., Principal Investigator — Samsun University; Mustafa Açıkgöz, Assoc. Prof, Study Director — Zonguldak Bulent Ecevit University; Nursena Ceylan, Principal Investigator — Zonguldak Bulent Ecevit University; Arzucan Toksal Uçar, Principal Investigator — Zonguldak Bulent Ecevit University
Locations (2):
- Turkey (Türkiye) (2):
  - Arzucan Toksal, Zonguldak
  - Zonguldak Bulent Ecevit University, Zonguldak